CLINICAL TRIAL: NCT02206074
Title: The Effect of Dietary Nitrate Supplementation on Ability of Individuals With Type 2 Diabetes to Perform Exercise
Acronym: Ex nit as
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Diabetes UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: CRF107; 12/SW/0118 (Other: NRES)
Record Dates: First submitted 2014-07-25; First posted 2014-08-01 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- T2DM (Active Comparator): Crossover design where participants will start in the Beetroot juice condition, and after a washout period, move into the other condition.
  Interventions: Dietary Supplement: Beetroot
- Placebo (Placebo Comparator): Crossover design where participants will start in the placebo condition, and after a washout period, move into the other condition.
  Interventions: Dietary Supplement: Beetroot

INTERVENTIONS:
Dietary Supplement: Beetroot
  Other Names: James Whites Drinks beetroot sports shot

SUMMARY:
The investigators are conducting a research study to see if increasing the amount of nitrate (a substance found in large quantities in certain vegetables) in the diet can increase the ability of individuals with Type 2 diabetes (T2D) to perform exercise. Some people with T2D find exercise more uncomfortable than individuals who do not have T2D. This may be explained by the experimental studies showing that T2D can result in reductions in the supply of oxygen to the muscles. Studies have also shown that for a given level of activity, individuals with T2D will be much closer to their maximum exercise capacity than healthy individuals. Dietary nitrate may have two important beneficial effects in individuals with T2D: 1) The effects of dietary nitrate on the responses to exercise may have a significant impact on the ability of individuals with Type 2 diabetes to perform daily tasks and exercise more comfortably and 2) experimental studies suggest that increased nitrate consumption has been shown to reduce the amount of oxygen required for a given level of exercise.

The investigators will recruit 60 individuals with T2D. These people will take part in a randomised crossover design study where they will be asked to drink normal beetroot juice (rich in nitrate) and nitrate depleted beetroot juice, prior to performing two different walking exercise tasks (a six minute walk and repeated, low intensity treadmill walking). This study aims to determine if dietary nitrate supplementation reduces the amount of oxygen required for a given level of exercise in individuals with T2D. To test brain function individuals will be asked to perform a standard computerised decision making task following consumption of the nitrate rich and nitrate depleted juices.

ELIGIBILITY:
Inclusion Criteria:

* patients with T2D (as defined by WHO) of at least 5 years duration between the ages of 35-75 will be invited.

Exclusion Criteria:

* patients with significant renal impairment (eGFR<30)
* uncontrolled hypertension
* BMI<25 or >35
* are taking regular organic nitrates, nicorandil, or thiazolidinidiones, or any medication which may interfere with data interpretation or safety
* who have had a myocardial infarction or cerebro-vascular event
* who smoke, or any other serious medical condition which would interfere with data interpretation or safety will be excluded from participation.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pulmonary gas exchange via MedGraphics CardiO2 Cardiopulmonary Diagnostic Systems | 3 x 6 minutes of gas exchange per participant, twice, 10-14 days apart
  Pulmonary gas exchange was measured during treadmill walking exercise (MedGraphics CardiO2 Cardiopulmonary Diagnostic Systems, St. Paul, MN, USA). Prior to each testing session the analysers were calibrated using known concentrations. The volume transducer was calibrated using a 3-litre syringe (Hans Rudolph, Kansas City, MO, USA). When we refer to the oxygen cost of exercise we are referring to end exercise oxygen uptake.

SECONDARY OUTCOMES:
Functional capacity measured by 6-Minute Walking Test (6MWT) | 6 minutes walking per participant per visit

CONTACTS AND LOCATIONS:
Overall Officials: Daryl Wilkerson, PhD, Principal Investigator — University of Exeter
Locations (1):
- Peninsula NIHr Exeter Clinical Research Facility, Exeter, Devon, United Kingdom

REFERENCES:
- [Derived] Shepherd AI, Gilchrist M, Winyard PG, Jones AM, Hallmann E, Kazimierczak R, Rembialkowska E, Benjamin N, Shore AC, Wilkerson DP. Effects of dietary nitrate supplementation on the oxygen cost of exercise and walking performance in individuals with type 2 diabetes: a randomized, double-blind, placebo-controlled crossover trial. Free Radic Biol Med. 2015 Sep;86:200-8. doi: 10.1016/j.freeradbiomed.2015.05.014. Epub 2015 May 18. PMID 25998421